CLINICAL TRIAL: NCT00841503
Title: A Double-Blind, Randomized, Controlled Study to Determine Buckwheat's Glucose Lowering Effects in Healthy Volunteers and Volunteers With Type 2 Diabetes
Brief Title: Exploring Buckwheat's Glucose Lowering Potential
Status: Completed | Type: Observational
Sponsor: St. Boniface Hospital (Other)
Collaborators: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr.Peter Zahradka, Professor, Department of Physiology, St. Boniface Hospital
Other Study IDs: buckwheat study
Record Dates: First submitted 2009-02-10; First posted 2009-02-11 (Estimated); Last update posted 2012-03-21 (Estimated); Status verified 2012-03

CONDITIONS: Type 2 Diabetes
Keywords: functional food study
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Glucose; Sweetening Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 12 healthy volunteers: Healthy volunteers are randomized to 1 of 4 products over 4 weekly visits: i)buckwheat crackers;ii)crackers without buckwheat; iii)oral glucose; iv) oral sugar substitute, followed by 7 days of buckwheat crackers.
  Interventions: Other: buckwheat, rice crackers, glucose, sugar substitute
- 12 Participants with Type 2 diabetes: Volunteers with type 2 diabetes are randomized to 1 of 4 products over 4 weekly visits: i)buckwheat crackers;ii)crackers without buckwheat; iii)oral glucose; iv) oral sugar substitute, followed by 7 days of buckwheat crackers.
  Interventions: Other: buckwheat, rice crackers, glucose, sugar substitute

INTERVENTIONS:
Other: buckwheat, rice crackers, glucose, sugar substitute — crackers contain equal amounts of available carbohydrates; 50 mls of oral solution for both glucose and Splenda

SUMMARY:
Bioactive components in buckwheat enhance insulin sensitivity in Type 2 diabetes by improving glucose uptake and utilization through a unique mechanism that operates independent of insulin.

DETAILED DESCRIPTION:
This is a single site, double-blind, randomized, controlled study designed to explore buckwheat's glucose lowering effects in healthy volunteers and volunteers with type 2 diabetes. A total of 24 volunteers consisting of 12 volunteers (healthy and diabetic) per group for both the acute and chronic phases of testing will be recruited through advertisement from the local community.

In the acute testing phase, volunteers (healthy and diabetic) will be asked to attend 4 visits one week apart for the duration of 3 hours per visit. A fasting blood sample will be collected at each visit. At each visit, all volunteers will consume in random order 1 of the following 4 products: i) crackers containing buckwheat; ii) crackers without buckwheat); iii) 50 mls of oral solution containing glucose; or iv) 50 mls of oral solution containing the sugar substitute Splenda. The crackers will contain equal amounts of available carbohydrates. Blood sampling will occur at 15, 30, 45, 60 minutes, and then every 60 minutes for the remainder of the visit. Sampling (pre and post product consumption) will measure insulin, glucose, and various incretins. Open venous access will be secured after the first sample has been obtained to minimize the number of needle pricks. Total amount of blood obtained will not exceed 30 mls per visit.

In the chronic testing phase, volunteers (healthy and diabetic) will receive the crackers containing buckwheat for consumption each day for 7 days. Prior to food consumption, a fasting blood sample will be obtained each day and a urine sample will be collected on Days 1, 3, and 7 to assess bioavailability of buckwheat compounds (concentrations in blood and urine), insulin and glucose. Sampling for a lipid profile (total cholesterol, LDL-cholesterol, HDL-cholesterol and triglycerides), liver (ALT), kidney (creatinine), adipose function (adipokines), various incretins, as well as inflammatory status (various cytokines) will be done on Day 1 and Day 7. Total amount of blood obtained will not exceed 30 mls per visit.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 to 70 years
* normal glycated hemoglobin (<6% healthy, <7.5% diabetic)
* absence of chronic conditions (except Type 2 diabetes)
* must be able to read and sign consent
* must be able to comply with protocol requirements

Exclusion Criteria:

* allergies to eggs, buckwheat, rice flour, or sugar substitutes (Splenda)
* acute or chronic conditions (except Type 2 diabetes)
* blood glucose >10mmol/L at beginning of test session
* medications that affect glycemic control

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 24 volunteers were recruited from the community; 12 healthy volunteers and 12 volunteers with Type 2 Diabetes
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2008-09; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
determine glucose-lowering potential of the buckwheat bioactive compound during acute phase testing in volunteers with Type 2 diabetes | 3 hour testing

SECONDARY OUTCOMES:
determine bioavailability of buckwheat bioactive compounds | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Peter C Zahradka, PhD, Principal Investigator — Canadian Centre for Agri-Food Research in Health & Medicine
Locations (1):
- I.H. Asper Clinical Research Institute, Winnipeg, Manitoba, Canada

REFERENCES:
- [Background] Kawa JM, Taylor CG, Przybylski R. Buckwheat concentrate reduces serum glucose in streptozotocin-diabetic rats. J Agric Food Chem. 2003 Dec 3;51(25):7287-91. doi: 10.1021/jf0302153. PMID 14640572
- [Background] Qureshi AA, Sami SA, Khan FA. Effects of stabilized rice bran, its soluble and fiber fractions on blood glucose levels and serum lipid parameters in humans with diabetes mellitus Types I and II. J Nutr Biochem. 2002 Mar;13(3):175-187. doi: 10.1016/s0955-2863(01)00211-x. PMID 11893482
- [Background] Knekt P, Kumpulainen J, Jarvinen R, Rissanen H, Heliovaara M, Reunanen A, Hakulinen T, Aromaa A. Flavonoid intake and risk of chronic diseases. Am J Clin Nutr. 2002 Sep;76(3):560-8. doi: 10.1093/ajcn/76.3.560. PMID 12198000
- [Background] Thompson LU, Robb P, Serraino M, Cheung F. Mammalian lignan production from various foods. Nutr Cancer. 1991;16(1):43-52. doi: 10.1080/01635589109514139. PMID 1656395
- [Background] Larner J, Huang LC, Schwartz CF, Oswald AS, Shen TY, Kinter M, Tang GZ, Zeller K. Rat liver insulin mediator which stimulates pyruvate dehydrogenase phosphate contains galactosamine and D-chiroinositol. Biochem Biophys Res Commun. 1988 Mar 30;151(3):1416-26. doi: 10.1016/s0006-291x(88)80520-5. PMID 2833261
- [Background] Larner J, Huang LC, Suzuki S, Tang G, Zhang C, Schwartz CF, Romero G, Luttrell L, Kennington AS. Insulin mediators and the control of pyruvate dehydrogenase complex. Ann N Y Acad Sci. 1989;573:297-305. doi: 10.1111/j.1749-6632.1989.tb15006.x. No abstract available. PMID 2517463
- [Background] Varela-Nieto I, Leon Y, Caro HN. Cell signalling by inositol phosphoglycans from different species. Comp Biochem Physiol B Biochem Mol Biol. 1996 Oct;115(2):223-41. doi: 10.1016/0305-0491(96)00087-9. PMID 8939003
- [Background] Field MC. Is there evidence for phospho-oligosaccharides as insulin mediators? Glycobiology. 1997 Mar;7(2):161-8. doi: 10.1093/glycob/7.2.161-d. No abstract available. PMID 9134421
- [Background] Jones DR, Varela-Nieto I. The role of glycosyl-phosphatidylinositol in signal transduction. Int J Biochem Cell Biol. 1998 Mar;30(3):313-26. doi: 10.1016/s1357-2725(97)00144-1. PMID 9611774
- [Background] Oku A, Ueta K, Arakawa K, Ishihara T, Nawano M, Kuronuma Y, Matsumoto M, Saito A, Tsujihara K, Anai M, Asano T, Kanai Y, Endou H. T-1095, an inhibitor of renal Na+-glucose cotransporters, may provide a novel approach to treating diabetes. Diabetes. 1999 Sep;48(9):1794-800. doi: 10.2337/diabetes.48.9.1794. PMID 10480610
- [Background] Adachi T, Yasuda K, Okamoto Y, Shihara N, Oku A, Ueta K, Kitamura K, Saito A, Iwakura I, Yamada Y, Yano H, Seino Y, Tsuda K. T-1095, a renal Na+-glucose transporter inhibitor, improves hyperglycemia in streptozotocin-induced diabetic rats. Metabolism. 2000 Aug;49(8):990-5. doi: 10.1053/meta.2000.7729. PMID 10954015
- [Background] Ueta K, Ishihara T, Matsumoto Y, Oku A, Nawano M, Fujita T, Saito A, Arakawa K. Long-term treatment with the Na+-glucose cotransporter inhibitor T-1095 causes sustained improvement in hyperglycemia and prevents diabetic neuropathy in Goto-Kakizaki Rats. Life Sci. 2005 Apr 22;76(23):2655-68. doi: 10.1016/j.lfs.2004.09.038. PMID 15792833
- [Background] Nawano M, Oku A, Ueta K, Umebayashi I, Ishirahara T, Arakawa K, Saito A, Anai M, Kikuchi M, Asano T. Hyperglycemia contributes insulin resistance in hepatic and adipose tissue but not skeletal muscle of ZDF rats. Am J Physiol Endocrinol Metab. 2000 Mar;278(3):E535-43. doi: 10.1152/ajpendo.2000.278.3.E535. PMID 10710509
- [Background] Skrabanja V, Liljeberg Elmstahl HG, Kreft I, Bjorck IM. Nutritional properties of starch in buckwheat products: studies in vitro and in vivo. J Agric Food Chem. 2001 Jan;49(1):490-6. doi: 10.1021/jf000779w. PMID 11170616
- [Background] Bray GA. Evaluation of obesity. Who are the obese? Postgrad Med. 2003 Dec;114(6):19-27, 38. doi: 10.3810/pgm.2003.12.1544. PMID 14689721
- [Background] Ball GD, McCargar LJ. Childhood obesity in Canada: a review of prevalence estimates and risk factors for cardiovascular diseases and type 2 diabetes. Can J Appl Physiol. 2003 Feb;28(1):117-40. doi: 10.1139/h03-010. PMID 12671200
- [Background] Lu C et al. (1992) Proceedings of the 5th International Symposium on Buckwheat; Lin R, Zhou M, Tao Y, Li J, Zhang, Z. Eds; Agriculture Publishing House: Beijing,China; pp 458-464.
- [Background] Wang J et al. (1992) Proceedings of the 5th International Symposium on Buckwheat; Lin R, Zhou M, Tao Y, Li J, Zhang, Z. Eds; Agriculture Publishing House: Beijing, China; pp 465-467.
- [Background] Horbowicz M & Obendorf RL. (1994) Seed Sci Res 4: 385-405.
- [Background] Obendorf RL, Steadman KJ, Fuller DJ, Horbowicz M, Lewis BA. Molecular structure of fagopyritol A1 (O-alpha-D-galactopyranosyl-(1 --> 3)-D-chiro-inositol) by NMR. Carbohydr Res. 2000 Oct 6;328(4):623-7. doi: 10.1016/s0008-6215(00)00133-6. PMID 11093720
- [Background] Steadman KJ, Burgoon MS, Schuster RL, Lewis BA, Edwardson SE, Obendorf RL. Fagopyritols, D-chiro-inositol, and other soluble carbohydrates in buckwheat seed milling fractions. J Agric Food Chem. 2000 Jul;48(7):2843-7. doi: 10.1021/jf990709t. PMID 10898633
- [Background] Steadman KJ, Fuller DJ, Obendorf RL. Purification and molecular structure of two digalactosyl D-chiro-inositols and two trigalactosyl D-chiro-inositols from buckwheat seeds. Carbohydr Res. 2001 Mar 9;331(1):19-25. doi: 10.1016/s0008-6215(00)00320-7. PMID 11284502
- [Background] Scheepers A, Joost HG, Schurmann A. The glucose transporter families SGLT and GLUT: molecular basis of normal and aberrant function. JPEN J Parenter Enteral Nutr. 2004 Sep-Oct;28(5):364-71. doi: 10.1177/0148607104028005364. PMID 15449578